CLINICAL TRIAL: NCT01392352
Title: HYPAZ: An Open-label Investigation Into Hypertension Induced by Pazopanib Therapy
Brief Title: HYPAZ: Hypertension Induced by Pazopanib
Acronym: HYPAZ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following DMC review, due to slow recruitment of evaluable patients.
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Duncan Jodrell, Professor Duncan Jodrell, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A091962; 2010-021613-23 (EudraCT Number)
Record Dates: First submitted 2011-06-30; First posted 2011-07-12 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Renal Cell Carcinoma; Soft Tissue Sarcoma; Glioblastoma; Ovarian Cancer; Cervical Cancer; Breast Cancer; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Pancreatic Cancer; Melanoma; Gastrointestinal Cancer
Keywords: pazopanib; hypertension; forearm blood flow
MeSH Terms: conditions — Carcinoma, Renal Cell; Sarcoma; Glioblastoma; Ovarian Neoplasms; Uterine Cervical Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Pancreatic Neoplasms; Melanoma; Gastrointestinal Neoplasms; Hypertension | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib (Experimental): Patients will receive 800mg (2 X 400mg tablets) of pazopanib, to be administered once daily orally for 12 weeks or until development of hypertension (defined as VHyp), whichever occurs first.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 2 x 400mg pazopanib tablets taken once daily for 12 weeks
  Other Names: Votrient

SUMMARY:
Pazopanib is a new cancer drug that works by limiting the growth of new blood vessels in tumours. About half of patients who take pazopanib develop high blood pressure (hypertension). This side effect can make patients have to reduce or stop their cancer treatment, and can cause other health problems. The aim of this study is to find out exactly how the drug causes high blood pressure.

DETAILED DESCRIPTION:
For this study, up to 52 patients with different cancer types will take pazopanib tablets for 12 weeks. They will visit the clinic every 1-2 weeks during treatment, and for a final safety check 4 weeks after stopping the drug (10 visits over 18 weeks).

At every visit, we will do a heart tracing, and check the patient's blood pressure and blood and urine chemicals (to check their health, and see if levels of these chemicals change). Patients will check their blood pressure at home every other day. They will also wear a blood pressure monitor for 24 hours on 3 occasions (during normal daily activities).

Patients will have 1 or 2 CT scans and 3 MRI scans during the study. On three occasions, a variety of specialised tests will measure how the patient's blood vessels are working.

Patients may choose to continue taking the drug after the 12 weeks of treatment, if their doctor feels it is appropriate.

Understanding how pazopanib causes high blood pressure will help us to advise doctors how to treat the high blood pressure effectively, so that patients can continue to take their cancer treatment safely. This research might also lead to the development of new cancer drugs in future, which do not cause this serious side effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up.
2. Patients with the following tumour types where VEGF inhibition would be appropriate therapy:

   a Renal cell carcinoma b Ovarian carcinoma with a rising CA-125, 2nd or subsequent lines c Ovarian carcinoma with residual disease after chemotherapy in the absence of rising CA-125, 2nd or subsequent lines d Cervical cancer, metastatic or recurrent, and progressing after conventional chemotherapy e Glioblastoma, progressing after conventional chemotherapy f Advanced or metastatic soft tissue sarcoma, residual disease post chemotherapy in the absence of progression, 2nd or subsequent lines g Advanced or metastatic soft tissue sarcoma progressing post conventional chemotherapy, 3rd or subsequent lines h Non-small cell lung cancer, 1st or subsequent lines i ErbB2 positive, advanced or metastatic breast cancer, 2nd or subsequent lines j Gemcitabine-refractory pancreatic cancer, 2nd or subsequent lines k Non-cutaneous (ocular or mucosal) melanoma and cutaneous melanoma any line l GI tract 2nd line residual disease or subsequent lines m Small Cell Lung cancer 3rd line n Other solid tumours in which anti-VEGF therapy is judged by the CI to be of possible clinical benefit
3. Measurable disease as per RECIST 1.1. A measurable lesion is defined as a lesion that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques. Patients with ovarian cancer or prostate cancer, where validated tumour markers (CA125 and PSA) are used clinically to monitor response, do not require measurable disease as per RECIST 1.1.
4. ECOG performance status 0 or 1.
5. Age ≥18 years.
6. Adequate organ system function
7. Female participant, or female partner of male participant, are of non-childbearing potential or agree to protocol-specified contraceptive measures

Exclusion Criteria:

1. Known hypertension (blood pressure >150/90 mmHg (± 2 mmHg, at investigator's discretion) at baseline
2. On anti-hypertensive therapy indicated for hypertension
3. History of any one or more of the following cardiovascular conditions within the last 6 months:

   a Cardiac angioplasty or stenting b Myocardial infarction c Unstable angina d Coronary artery bypass graft surgery e Peripheral vascular disease or Raynaud's phenomenon f Cerebrovascular accident (CVA) including transient ischaemic attack (TIA), g Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
4. Hypersensitivity to agents used in forearm blood flow studies (acetylcholine, sodium nitroprusside, L-NMMA)
5. Difficult upper limb arterial access (as assessed by an easily palpable brachial artery)
6. Anticoagulant therapy (warfarin). (Subcutaneous heparin is allowed but will need to be omitted on visits V2, V3 and VHyp).
7. Pregnant or lactating female
8. History or clinical evidence of active central nervous system (CNS) metastases.
9. Clinically significant gastrointestinal abnormalities that may increase the risk for GI bleeding
10. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
11. Presence of uncontrolled infection
12. Corrected QT interval (QTc) > 480 msecs using Bazett's formula
13. History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
14. Prior major surgery or trauma within 28 days prior to first dose and/or presence of any non-healing wound, fracture, or ulcer.
15. Evidence of active bleeding or bleeding diathesis
16. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.

    Note: Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, the presence of a tumour that is touching, but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions).

    i) Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed.

    ii) Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.
17. Significant haemoptysis within 8 weeks prior to first dose of pazopanib (≥½ teaspoon of red blood within 8 weeks before first dose of study drug).
18. Any serious and/or pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent, or compliance to study procedures.
19. Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib and for the duration of the study.
20. Treatment with any of the following anti-cancer therapies:

    a radiation therapy (single fraction radiotherapy for pain control is allowed in this period and when on study), surgery or tumour embolization within 14 days prior to the first dose of pazopanib OR b chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib c pazopanib or other antiangiogenic treatment (e.g. bevacizumab) within the past 12 weeks.
21. Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment.
22. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
23. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in endothelial dependent function | Measured over 12 weeks, or at the onset of hypertension whichever occurs first

SECONDARY OUTCOMES:
Change in endothelial independent function | Measured over 12 weeks, or at onset of hypertension, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Duncan I Jodrell, Principal Investigator — University of Cambridge; honorary contract with Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Maki-Petaja KM, McGeoch A, Yang LL, Hubsch A, McEniery CM, Meyer PAR, Mir F, Gajendragadkar P, Ramenatte N, Anandappa G, Santos Franco S, Bond SJ, Schonlieb CB, Boink Y, Brune C, Wilkinson IB, Jodrell DI, Cheriyan J. Mechanisms Underlying Vascular Endothelial Growth Factor Receptor Inhibition-Induced Hypertension: The HYPAZ Trial. Hypertension. 2021 May 5;77(5):1591-1599. doi: 10.1161/HYPERTENSIONAHA.120.16454. Epub 2021 Mar 29. PMID 33775123